CLINICAL TRIAL: NCT02852616
Title: Progression and Remittance of Traumatic Stress-related Symptoms During and After Narrative Exposure Therapy
Brief Title: Trajectories of Psychopathology in Response to NET
Acronym: TOP-NET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Elbert, Professor for Clinical Psychology and Behavioural Neuroscience, University of Konstanz
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERC-2012-AdG 323977 NET-Course
Record Dates: First submitted 2016-06-01; First posted 2016-08-02 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2018-10

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: Course; Posttraumatic Stress Disorder; Narrative Exposure Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Narrative Exposure Therapy (Active Comparator): Participants with a PTSD diagnosis
  Interventions: Behavioral: Narrative Exposure Therapy
- no / standard treatment (No Intervention): Participants with a PTSD diagnosis / other mental health problems / no mental health problems

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy — 8 - 15 sessions: 1 lifeline session, 5 - 12 sessions narrative exposure, 1-2 sessions of future-oriented counselling
  Other Names: NET
  Arms: Narrative Exposure Therapy

SUMMARY:
Narrative Exposure Therapy (NET) has been proven to be effective in the treatment of Posttraumatic Stress Disorder (PTSD) and trauma-related depression in more than a dozen controlled clinical trials. Symptom reduction was greatest during long-term follow-ups after the completion of the therapy.

In the current study, we will investigate the progression of PTSD symptoms and emotional stress before, during and after therapy. After a semi-structured interview all participants will be asked to report in monthly telephone interviews their core symptoms. Structured interviews after 6 and 12 months are used to validate the outcome. A convenience sample of individuals with a PTSD will be offered participation in the study.

DETAILED DESCRIPTION:
Participants will be recruited through the Center of Excellence for Psychotraumatology, University of Konstanz, with focus on refugees. All of them (approx. 100) will receive a structured interview and a detailed diagnosis. The interview includes questions about sociodemography, traumatic events, PTSD and depression symptomatology. Individuals with a PTSD diagnosis (up to 30) will be offered a Narrative Exposure Therapy (NET).

Irrespective of treatment and diagnosis, respondents are asked to participate in monthly telephone interviews assessing trauma-related and emotional distress and changes in life. Interviews assessing PTSD, depression symptoms and emotional distress will be conducted 6 and 12 months after the initial interview.

In addition, participants receiving NET will rate their PTSD symptoms and functionality prior to each therapy session.

ELIGIBILITY:
Inclusion Criteria:

* For treatment group: PTSD diagnosis (DSM-IV or V)
* For non-treatment group: none

Exclusion Criteria:

* Acute psychosis
* Cerebro-organic disease
* Acute drug or alcohol intoxication
* Already receiving another psychotherapy
* Anti-epileptic drugs at baseline

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in the progression of PTSD symptoms (PCL-5) | baseline, 3 and 6 months follow-up
  PTSD symptoms are measured with the PTSD Checklist - 5 (PCL-5; Weathers, Litz, et al., 2013)

SECONDARY OUTCOMES:
Change in the progression of emotional distress symptoms (RHS-15) | up to 1 year
  Emotional distress symptoms are measured with the Refugee Health Screener - 15 (RHS-15; Hollifield, et al., 2013)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Elbert, Prof. Dr., Principal Investigator — University of Konstanz
Locations (1):
- University of Konstanz, Konstanz, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaltenbach E, Hermenau K, Schauer M, Dohrmann K, Elbert T, Schalinski I. Trajectories of posttraumatic stress symptoms during and after Narrative Exposure Therapy (NET) in refugees. BMC Psychiatry. 2020 Jun 17;20(1):312. doi: 10.1186/s12888-020-02720-y. PMID 32552778